CLINICAL TRIAL: NCT01012115
Title: Temporal Behavior of Coagulation Factors,Cytokines and Tissue Injury Markers in Sepsis: Validation of Extracellular Histones
Brief Title: Coagulation Factors, Cytokines and Tissue Injury Markers in Sepsis
Acronym: Histone
Status: Completed | Type: Observational
Sponsor: University of Oklahoma (Other)
Collaborators: Oklahoma Medical Research Foundation (Other)
Responsible Party: Principal Investigator, Gary Kinasewitz, Principal Investigator, University of Oklahoma
Other Study IDs: 14849
Record Dates: First submitted 2009-11-09; First posted 2009-11-11 (Estimated); Last update posted 2012-04-09 (Estimated); Status verified 2012-04

CONDITIONS: Sepsis
Keywords: Histones; organ failure; sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
In an effort to better understand the interaction between the different mediators, the investigators propose to examine the time course of mediators, the indexes of organ injury and the coagulation cascade.

DETAILED DESCRIPTION:
All patients admitted to the ICU (Including VA Medical Center, University Hospital and Presbyterian hospital) will be screened for enrollment in the study. Patients who have the diagnosis of sepsis will be asked to volunteer. We will match sepsis patients with other ICU patients without the diagnosis of sepsis. The latter will also be asked to volunteer.

Patients will be stratified into three groups:

* Sepsis
* SIRS of non-septic origin
* Other ICU patients

Routine laboratory data and clinical data (see flow sheet) will be collected. The plasma or serum will be frozen separately until the target number of patients is met. Measurements of inflammatory mediators and other cytokines/injury markers will be carried out at that point.

ELIGIBILITY:
Inclusion Criteria:

* Admission to the ICU

Exclusion Criteria:

* No blood draws scheduled
* Hemoglobin level < 6.5 gm/dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the ICU with suspected or proven sepsis.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2009-10; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary T Kinasewitz, MD, Principal Investigator — OU Health Sciences Center
Locations (2):
- United States (2):
  - OU Medical Center, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center, Oklahoma City, Oklahoma